CLINICAL TRIAL: NCT03054610
Title: Therapeutic Effect of Botulinum Toxin A for the Treatment of Plantar Fasciitis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR15-001
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Plantar Fascitis; Botulinum Toxins, Type A
Keywords: plantar fascitis; Botulinum toxin A; Betamethason Sodium Phosphate; infiltration; plantar fascia
MeSH Terms: interventions — betamethasone sodium phosphate; betamethasone acetate phosphate; Ropivacaine; Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): 5 ml of local anesthetic (ropivacaine 7.5%)
  Interventions: Drug: Ropivacaine
- Steroid (Active Comparator): 1ml of steroid Betamethason Sodium Phosphate (Celestone®) and local anesthetic (ropivacaine 7.5%)
  Interventions: Drug: Betamethason Sodium Phosphate; Drug: Ropivacaine
- BTX-A (Experimental): 200U Botulinum Toxins, Type A
  Interventions: Drug: Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate
  Other Names: Celestone Soluspan
  Arms: Steroid
Drug: Ropivacaine
  Other Names: Ropiconest
  Arms: Control; Steroid
Drug: Botulinum Toxins, Type A
  Other Names: Dysport
  Arms: BTX-A

SUMMARY:
Plantar fasciitis is the most common cause of plantar heel pain and is commonly present in people 40 years of age or older, overweight, sedentary or with intense physical activity. It is caused by the over-stretching of the plantar fascia, which is a band of connective tissue that extends to the base of the phalanges. This produces micro-tears more commonly in its origin in the medial tuberosity of the calcaneus which causes an inflammatory process and pain. This pain usually occurs when the person gets up in the morning after sleeping or after sitting for a long time. That is when the fascia is stretched after being in a contraction position.

There are a great variety of treatments for this pathology, of these, one of the most common is the use of intralesional steroids, which a weighing that reduces symptomatology in many cases also has undesirable effects such as subcutaneous fat atrophy, rupture of the plantar fascia, peripheral nerve injury, muscle damage and stress fractures. Other treatments are extracorporeal shock waves, application of platelet-rich plasma and application of botulinum toxin A intralesional. All of them are accompanied by insoles, night splints and stretching exercises of the Achilles tendon and the plantar fascia.

Recent studies have shown that the application of botulinum toxin A intralesional in patients with plantar fasciitis helps to improve the symptomatology to decrease pain in both intensity and presentation time. Decreased inflammation of the plantar fascia has also been demonstrated. This is the sale of the usual form of action of the botulinum toxin, which is applied regularly in the muscles to block the release of acetylcholine in the neuromuscular plaque and obtain its relaxation and not directly in the pain points. We believe that the botulinum toxin can be applied intralesional currently, since there is information that the toxin has analgesic and anti-inflammatory effect and not just muscle relaxation.

The aim of our work demonstrate that the use of botulinum toxin A and intralesional stretching exercises is superior to intralesional steroids and stretching trying to establish a safer and less painful therapy avoiding complications prior to the application of steroid application.

DETAILED DESCRIPTION:
Plantar fasciitis represents the most frequent cause of chronic heel pain, usually occurs in patients 40 years or older, overweight, sedentary or with intense physical activity.

The plantar fascia function is to prevent foot collapse by its anatomical orientation and by its tensile forces; It originates at the base of the calcaneus and extends distally to the phalanges. The plantar fascia stretching prevents the displacement of the calcaneus and the metatarsals and maintains the medial longitudinal arch. Simulates a cable attached to the calcaneus and metatarsophalangeal joints. The windlass mechanism described by Hicks, for the action of the plantar fascia is usually explained when a dorsiflexion of the fingers occurs, this leads to an effective shortening of the length of the plantar fascia causing an elevation of the arch. The extension of the fingers increases the arch of tension with the metatarsophalangeal joint as axis or anchor point. The shortening of the plantar fascia resulting from the dorsiflexion of the hallux is the essence of the windlass mechanism. When a fasciotomy is performed, this mechanism is lost, decreasing the stability of the arch and this does not allow a phase of stable terminal stay.

Historically the development of plantar fasciitis is attributed to biomechanical defects such as hyperpronation, this contributes to excesive mobility of the foot, which increases the stress applied to the musculofascial structures and soft tissue through an elongation of plantar fascia. There are other studies that have shown that one of the main factors for the appearance of this disease is the mechanical overload and it has been reported that the tension necessary for the rupture of the windlass mechanism ranges from 1.4 to 3.4 of the body weight of the subject.

There is a great variety of therapies reported for the treatment of this pathology, intralesional application of steroids, platelet-rich plasma, intralesional botulinum toxin A, treatments such as extracorporeal shock waves, all of which are assisted by stretching excercises of the gastrocnemius and sole muscles or stretching of the plantar fascia.

The clinical use of botulinum toxin A has expanded beyond the original indications by its effects on cholinergic neurons. The increased interest in the potential role to treat conditions of chronic pain is partially based on the effects of the toxin on the modulation of the release of substance P, on the calcitonin-related gene peptide and glutamate. On the other hand, the toxin has shown its effect on the inhibition of inflamatory pain and on the release of neurotransmitters from primary sensory neurons in a rat model. It also inhibits peripheral sensitization, which leads to an indirect decrease in central sensitization. It is unclear whether the treatment of chronic plantar fasciitis with botulinum toxin A works by causing muscle paralysis or by analgesic anti-inflamatory effects or by both mechanisms. A combined effect, induction of paresia of the muscles originating in the medial calcaneus process and direct analgesia due to analgesic anti-inflamatory properties.

We performed a previous study, where we compared the use of botulinum toxin A against intralesional steroids; The application of botulinum toxin A was performed in the twin and sole muscle wombs, while dexamethasone was applied in the area of greatest fascia pain. Patients who received botulinum toxin had a faster and more sustained improvement than patients who received steroids.

Another common form of treatment for plantar fasciitis is the application of intralesional steroids; however, there are reports of complications associated with these drugs and one of the main ones is the rupture of the plantar fascia, which ranges from 2.4% to 5.7% ; Despite pain relief due to rupture, many patients have other associated complications such as lateral plantar nerve dysfunction, stress fractures, among others, mainly after 2 applications.

Objective and originality: The aim of our study is to demonstrate that the use of botulinum toxin A for the treatment of plantar fasciitis is superior to treatment with intralesional steroids. We try to establish a safer and less painful treatment therapy for the patient, since the use of steroids is associated with complications. We believe that the botulinum toxin A can also be applied intralesional, since there is information that indicates that this toxin has analgesic and anti-inflammatory effect in its local application and not only by the action of muscle relaxation by blocking the release of acetylcholine at the neuromuscular junctions.

General objective:

To assess the therapeutic effect of botulinum toxin A in patients diagnosed with plantar fasciitis.

Hypothesis:

The application of botulinum toxin A presents better results in the treatment of plantar fascitis than the use of intralesional steroids.

Material and Methods:

All patients who are recruited for the study will be explained regarding the treatment protocol, and will also sign informed consent prior to inclusion in the study. Measurement of the plantar fascia using ultrasound and measurement of ranges of movement of ankle flexion, as well as measuring and weighing patients to know their body mass index. They will be randomized into one of three treatment groups. Group 1 (control) treatment with 5 ml of anesthetic (Ropivacaine 7.5%), Group 2 (steroids) application of 1ml of Betamethasone plus 3 ml of local anesthetic and Group 3 (botulinum toxin A) 250 U, in the insertion zone of the plantar fascia. All patients will receive a detailed explanation of the stretching exercises of the plantar fascia, as well as their frequency and duration. Afterwards, the patients will be evaluated by a blinded investigator, at 2 weeks, 1 month, 3 months and 6 months after infiltration; evaluation scales will be applied: Visual Analogue Scale (EVA), Maryland Foot & Ankle Score, Foot & Ankle Outcome Score (AOFAS), Foot & Ankle Disability Index (FADI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain in the heel at the insertion of the plantar fascia in the posteroinferior tuberosity of the calcaneus.
* Patients who agreed to be part of the study and signed informed consent.
* Patients older than 18 years.
* Patients with two or more weeks of evolution.

Exclusion Criteria:

* Patients with another associated pathology such as knee or ankle dysfunction, osteoarthritis, rheumatoid arthritis, ankylosing spondylitis, etc.
* Neurological abnormalities: mental retardation or some psychiatric abnormality.
* Pregnant patients.
* Previous surgery on the heel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Disability Index | 6 months
  We decided to include the FADI score because this type of pathology occurs in patients with sports activity and often causes disability in them, Values activities such as standing, walking on flat or uneven surfaces, inclined planes, time without discomfort while walking, and includes a module where sports activities are valued. Also it counts on an evaluation of the pain in foot and ankle. The best result obtained is 136 points.

SECONDARY OUTCOMES:
Maryland Foot Score | 6 months
  Is divided into several sections where pain is assessed, giving 45 points when there is no pain and 0 when there is inability to work, a function that is divided into two sections, walking and daily activities; And a section that evaluates the shape of the foot, the best score is 100, which means that there is no problem with the foot, and the lowest score is 0.
Ankle-Hindfoot Scale | 6 months
  American Foot and Ankle Orthopedic Society
Visual Analogue scale | 6 months
  Values the pain on a numerical scale of 0-10, where 0 means no pain and 10 greater degree of pain experienced by the patient, it is also complemented by a color scale, where green is equal to painless and red is the more intense pain the patient has had.
Measurement of the plantar fascia using ultrasound | 6 months
  Measure the thickness of the plantar fascia at the beginning and end of the protocol, placing the transducer at the insertion site of the plantar fascia.
Body Mass Index | 15 minutes
  Measure height and weight of patients at the beginning of the protocol.
Measure degrees of dorsiflexion | 6 months
  Use a goniometer as a tool to measure degrees of dorsiflexion.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irving DB, Cook JL, Menz HB. Factors associated with chronic plantar heel pain: a systematic review. J Sci Med Sport. 2006 May;9(1-2):11-22; discussion 23-4. doi: 10.1016/j.jsams.2006.02.004. Epub 2006 Apr 3. PMID 16584917
- [Background] Taunton JE, Ryan MB, Clement DB, McKenzie DC, Lloyd-Smith DR, Zumbo BD. A retrospective case-control analysis of 2002 running injuries. Br J Sports Med. 2002 Apr;36(2):95-101. doi: 10.1136/bjsm.36.2.95. PMID 11916889
- [Background] May TJ, Judy TA, Conti M, Cowan JE. Current treatment of plantar fasciitis. Curr Sports Med Rep. 2002 Oct;1(5):278-84. doi: 10.1249/00149619-200210000-00005. PMID 12831690
- [Background] Kim C, Cashdollar MR, Mendicino RW, Catanzariti AR, Fuge L. Incidence of plantar fascia ruptures following corticosteroid injection. Foot Ankle Spec. 2010 Dec;3(6):335-7. doi: 10.1177/1938640010378530. Epub 2010 Sep 3. PMID 20817847
- [Background] Acevedo JI, Beskin JL. Complications of plantar fascia rupture associated with corticosteroid injection. Foot Ankle Int. 1998 Feb;19(2):91-7. doi: 10.1177/107110079801900207. PMID 9498581
- [Background] Glazer JL. An approach to the diagnosis and treatment of plantar fasciitis. Phys Sportsmed. 2009 Jun;37(2):74-9. doi: 10.3810/psm.2009.06.1712. PMID 20048512
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Rompe JD, Cacchio A, Weil L Jr, Furia JP, Haist J, Reiners V, Schmitz C, Maffulli N. Plantar fascia-specific stretching versus radial shock-wave therapy as initial treatment of plantar fasciopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2514-22. doi: 10.2106/JBJS.I.01651. PMID 21048171
- [Background] Soomekh DJ. Current concepts for the use of platelet-rich plasma in the foot and ankle. Clin Podiatr Med Surg. 2011 Jan;28(1):155-70. doi: 10.1016/j.cpm.2010.09.001. PMID 21276524
- [Background] Digiovanni BF, Nawoczenski DA, Malay DP, Graci PA, Williams TT, Wilding GE, Baumhauer JF. Plantar fascia-specific stretching exercise improves outcomes in patients with chronic plantar fasciitis. A prospective clinical trial with two-year follow-up. J Bone Joint Surg Am. 2006 Aug;88(8):1775-81. doi: 10.2106/JBJS.E.01281. PMID 16882901
- [Background] Tsai WC, Hsu CC, Chen CP, Chen MJ, Yu TY, Chen YJ. Plantar fasciitis treated with local steroid injection: comparison between sonographic and palpation guidance. J Clin Ultrasound. 2006 Jan;34(1):12-6. doi: 10.1002/jcu.20177. PMID 16353228
- [Background] Placzek R, Deuretzbacher G, Meiss AL. Treatment of chronic plantar fasciitis with Botulinum toxin A: preliminary clinical results. Clin J Pain. 2006 Feb;22(2):190-2. doi: 10.1097/01.ajp.0000169674.34191.0e. PMID 16428954
- [Background] Seyler TM, Smith BP, Marker DR, Ma J, Shen J, Smith TL, Mont MA, Kolaski K, Koman LA. Botulinum neurotoxin as a therapeutic modality in orthopaedic surgery: more than twenty years of experience. J Bone Joint Surg Am. 2008 Nov;90 Suppl 4:133-45. doi: 10.2106/JBJS.H.00901. No abstract available. PMID 18984726
- [Background] Elizondo-Rodriguez J, Araujo-Lopez Y, Moreno-Gonzalez JA, Cardenas-Estrada E, Mendoza-Lemus O, Acosta-Olivo C. A comparison of botulinum toxin a and intralesional steroids for the treatment of plantar fasciitis: a randomized, double-blinded study. Foot Ankle Int. 2013 Jan;34(1):8-14. doi: 10.1177/1071100712460215. PMID 23386757